CLINICAL TRIAL: NCT01275768
Title: A Double Blind, Randomized Controlled Prospective Trial of Endo-biliary Radio-frequency Ablation for Maintenance of Metal Stent Patency in Patients With Malignant Obstructive Jaundice
Brief Title: Role of Endoscopic RFA in Prolonging the Patency of Metal Stents in Patients With Malignant Obstructive Jaundice
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Dr. D. Nageshwar Reddy, Chairman, Asian Institute of Gastroenterology
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIG-GI-201101
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2011-01-14 (Estimated); Status verified 2011-01

CONDITIONS: Jaundice Extrahepatic Obstructive; Disorder of Bile Duct Stent
Keywords: radio-frequency ablation; Malignant jaundice

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): Insertion and activation of the endo-biliary RF catheter at the site of the stricture before insertion of a Self-expandable Metal Stent (SEMS)
  Interventions: Procedure: Endoscopic radio-frequency ablation
- Control arm (Placebo Comparator): Insertion and sham activation of the endo-biliary RF catheter at the site of the stricture before insertion of a SEMS
  Interventions: Procedure: Endoscopic radio-frequency ablation

INTERVENTIONS:
Procedure: Endoscopic radio-frequency ablation — Endobiliary radiofrequency catheter is 8Fr in diameter and can easily be passed over a 0.035 guide wire through the biopsy channel of a duodenoscope at the time of endoscopic retrograde cholangiography (ERC). Its use in the biliary system was heralded by animal experiments following which power settings of 7-10 Watts for 2 minutes were found to provide adequate ablation. The ablation results in charring of the tumor and this is expected to enhance the patency of SEMS

SUMMARY:
Patients with malignant obstructive jaundice (cancer of head of pancreas and cholangiocarcinoma) generally have a very poor prognosis with less than 20% patients having resectable disease at presentation. These patients also have a very poor quality of life with a life expectancy of 6-8 months. Jaundice associated with pruritus, poor appetite, malabsorption and loss of weight and cholangitis is the most common and troublesome problem. Placement of metallic stents has been the standard of care for patients with unresectable disease. However, about 50% of these stents get blocked in 6-8 months. Use of endoscopic Radio-frequency Ablation (RFA) prior to placement of metal stents may increase the patency of these stents

DETAILED DESCRIPTION:
We assume that application of endobiliary RFA to the malignant stricture which results in considerable charring of the tumor would result in prolongation of Self-expandable metal Stent (SEMS) patency by decreasing tumor in-growth and overgrowth. It is further speculated that prolonged stent patency will improve the quality of life of these patients, prevent cholangitis and optimize chemotherapy. A further outcome may be an improvement in the survival.

The research questions which we intend to answer through this trial would be:

1. Does application of prior endo-biliary radiofrequency affect patency of SEMS?
2. What are the complications associated with the use of endo-biliary RFA?
3. Does endo-biliary RFA with immediate placement of SEMS improve patient survival?
4. Is there any improvement in the quality of life of the patient with the combined use of endo-biliary RFA and SEMS?

Study protocol:

The study design is a double blind, sham operated, randomized controlled trial.

Inclusion criteria:

1. Patients: Clinical data and investigations suggestive of unresectable malignant bile duct obstruction. All patients will be discussed at the hepato-biliary multidisciplinary meeting which should come to a unanimous decision on tumor unresectability.
2. Age more than 18 years
3. Histologically/ Cytologically confirmed malignancy
4. Informed consent: The patient should voluntarily agree to participation and randomization. Oral and written information about the nature of the trial will be given to all patients considered for inclusion.

Exclusion Criteria:

1. Informed consent not obtained or withdrawn
2. Extremely poor general condition not amenable for conscious sedation used for Endoscopic retrograde Cholangiography (ERC)
3. Candidate suitable for surgical resection
4. Klatskin type 4 tumor
5. Previous biliary intervention such as plastic stent insertion for more than 1 month
6. Any other contra-indication to ERC

Randomization:

After obtaining an informed consent and satisfying the inclusion criteria, the patients will be randomized to one of the following two arms using computer generated randomization blocks. The operator and the patient will be blinded to use of RFA

1. Experimental arm: Insertion and activation of the endo-biliary RF catheter at the site of the stricture before insertion of a SEMS
2. Control arm: Insertion and sham activation of the endo-biliary RF catheter at the site of the stricture before insertion of a SEMS.

All patients will get the same SEMS with variable lengths (depending on the stricture size) to maintain uniformity. Endoscopic sphincterotomy will be performed in all patients prior to endo-biliary RF application and SEMS insertion. Opacification of the cystic duct and whether the endo-biliary RFA catheter was placed at the cystic duct opening will be recorded.

Data Collection:

Baseline data will be collected by an advanced endoscopy fellow and will include age, gender, WHO performance score, presence of gall bladder or gall stones, primary tumor type and stage, baseline liver function test, adjuvant chemo/radiotherapy

After discharge from the hospital, the patients will be followed up in the clinic at 1 week, 1 month, 3 months, 6 months, 9 months and 12 months. At each visit, a detailed clinical history, examination, adverse events, adjuvant therapy and liver function tests will be carried out. Patients will be assessed according to the World Health Organization performance classification.

WHO score

* 0 - Asymptomatic (Fully active, able to carry on all predisease activities without restriction)
* 1 - Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature. For example, light housework, office work)
* 2 - Symptomatic, <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours)
* 3 - Symptomatic, >50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours)
* 4 - Bedbound (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair)
* 5 - Death All patients will be referred for an oncological opinion for palliative chemotherapy. The patients and their care-givers will be told about symptoms of cholangitis and stent obstruction and will be asked to contact the hospital immediately in such cases. In the event of a confirmed SEMS occlusion, either a new SEMS or a plastic stent will be placed depending on the patient's prognosis.

End points:

1. Stent occlusion:

   1. Cholangitis
   2. or serum bilirubin > 3mg/dL with a previously normal bilirubin or above the baseline.
   3. Any clinical jaundice should be confirmed as being caused by stent occlusion by imaging or ERC
2. Death
3. Uneventful follow-up for 12 months

Evaluation:

The primary aim will be to compare the two groups for duration of stent patency.

The secondary aims will be:

1. To study any complications attributable to endo-biliary RFA
2. To study if there is any improvement in patient survival
3. To study if there is any improvement in patient's quality of life

Statistics:

We assume that the metal stent patency will improve from 50% to 80% at 6-8 months. With a 80% power and alpha error of 5%, we will need 43 patients in each arm. The Fisher exact test will be used to evaluate any differences in the patient distribution. The Student unpaired t test will be used to compare the laboratory tests, age and sex. Cumulative stent patency and patient survival will be estimated using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

1. Patients: Clinical data and investigations suggestive of unresectable malignant bile duct obstruction. All patients will be discussed at the hepato-biliary multidisciplinary meeting which should come to a unanimous decision on tumor unresectability.
2. Age more than 18 years
3. Histologically/ Cytologically confirmed malignancy
4. Informed consent: The patient should voluntarily agree to participation and randomization. Oral and written information about the nature of the trial will be given to all patients considered for inclusion.

Exclusion Criteria:

1. Informed consent not obtained or withdrawn
2. Extremely poor general condition not amenable for conscious sedation used for ERC
3. Candidate suitable for surgical resection
4. Klatskin type 4 tumor
5. Previous biliary intervention such as plastic stent insertion for more than 1 month
6. Any other contra-indication to ERC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Time to stent occlusion | 12 months
  Defined by a. Cholangitis b. or serum bilirubin > 3mg/dL with a previously normal bilirubin or above the baseline.
  c. Any clinical jaundice should be confirmed as being caused by stent occlusion by imaging or ERC

SECONDARY OUTCOMES:
Death | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: D. Nageshwar Reddy, DM, Study Director — Asian Institute of Gastroenterology
Locations (1):
- D. Nageshwar Reddy, Hyderabad, Andhra Pradesh, India